CLINICAL TRIAL: NCT03140163
Title: Screening for Pneumonia: A Comparison of Ultra Low Dose Chest CT and Conventional Chest Radiography
Brief Title: Screening for Pneumonia: A Comparison of Ultra Low Dose Chest CT [ULD-CT] and Conventional Chest Radiography [CXR]
Acronym: ULTRACHEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METC161004
Record Dates: First submitted 2016-09-16; First posted 2017-05-04 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subjects suffering from pneumonia (Experimental): CXR ULD-CT
  Interventions: Radiation: ULD-CT; Radiation: CXR

INTERVENTIONS:
Radiation: ULD-CT — Siemens Healthcare SOMATOM FORCE Ultra Low Dose chest CT
  Other Names: Ultra Low Dose chest CT
Radiation: CXR — Conventional chest radiograph
  Other Names: Conventional chest X ray

SUMMARY:
The ULTRACHEST study will be a prospective clinical diagnostic performance study with primary objective to establish device diagnostic clinical performance of Ultra Low Dose CT (ULD-CT) in order to prove it is more accurate in detecting pneumonia when comparing to standard conventional chest radiography.

DETAILED DESCRIPTION:
* 200 subjects
* Each subject will undergo CXR and ULD-CT at the same day.
* Subjects subdivided into 3 groups [high, moderate and low risk], based on a laboratory finding(CRP), symptoms and physical examination.
* 3 different thoracic radiologist will judge the scans on existence of consolidation. Consolidation will be expressed as binary outcomes (Yes or No consolidation)
* Radiologist will be blinded for subjects demographic data.
* All radiologist have to score how confidence they were on the finding of consolidation[5point likert].
* The investigators will perform a McNemar's test for evaluation. A two sided p-value of less than 0.05 will be considered to be statistically significant.
* Inter-observer variability will be evaluated by using a Fleiss Kappa test.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from pneumonia and referred by their GP

Exclusion Criteria:

* Younger than 18
* Known pregnancy
* Not able to sign the Informed Consent document
* If not willing to be informed about additional findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Three different radiologists will be asked to fill in a questionaire on whether or not there is presence of consolidation (yes/no) on both ULD-CT, as well as on CXR. | 2 years
  * 3 different thoracic radiologist will judge the scans on existence of consolidation. Consolidation will be expressed as binary outcomes (Yes or No consolidation)
  * Radiologist will be blinded for subjects demographic data.
Risk assessment of having a pneumonia for each subject | 2 year
  Subjects will be subdivided into 3 groups [high, moderate and low risk], based on a laboratory finding(CRP).
  * CRP levels lower than 20mg/L > low risk
  * CRP levels between 20 and 100mg/l > medium risk
  * CRP levels higher than 100mg/l > high risk
5 point likert scale to evaluate the "level of confidence" of each radiologist | 2 year
  - As described in "outcome 1" the radiologist judges the scans on existence of consolidation. After each judgement the radiologists has to fill in a questionaire [5 point likert scale] to score their level of confidence on the finding on whether or not they saw consolidation on the scan.

SECONDARY OUTCOMES:
All 3 radiologist will be asked to write down on paper if they see an additional finding on either the ULD-CT or CXR | 2 years
  Three different thoracic radiologist will judge the scans and fill in a questionaire if they see any additional finding (Yes/No).
In case the radiologist observes an additional finding, the radiologist has to fill in a questionaire on paper what kind of additional finding was seen: | 2 year
  In case they see an additional finding, they have to fill in what kind of additional finding the have seen and write it down in the questionaire.
  Example:
  [tumoral mass; pleural effusion; atelectasis; lymph nodules].
  - Additional findings will be subdivided in: atelectasis, pleural effusion, tree in bud, lymph nodes or tumoral mass.
Reporting the total number of observed additional findings for each modality [ULD-CT and CXR], based on the above mentioned questionaires | 2 year
  All additional findings will be presented in a table.
  for example:
  Number of subjects with additional finding of atelectasis:
  * ULD-CT (40 ULD-CT scans with atelectasis out of 100)
  * CXR (25 CXR radiographs with atelectasis out of 100)
  Number of subjects with additional finding of tumoral mass:
  * ULD-CT (2 ULD-CT scans with tumoral mass out of 100)
  * CXR (1 CXR radiographs with tumoral mass out of 100)
  Number of subjects with additional finding of pleural effusion:
  * ULD-CT (15 ULD-CT scans with pleural effusion out of 100)
  * CXR (33 CXR radiographs with pleural effusion out of 100)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Das, Dr, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- MUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No